CLINICAL TRIAL: NCT06719102
Title: Mothers and CareGivers Investing in Children: MAGIC 2.0
Brief Title: Mothers and CareGivers Investing in Children Study 2.0
Acronym: MAGIC 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Elizabeth Widen, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UT Austin IRB#STUDY00005620
Record Dates: First submitted 2024-10-23; First posted 2024-12-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Childhood Obesity Prevention; Parenting Behavior; Infant Growth
Keywords: Parenting; Infant Feeding; Infant Nutrition; Prevention; Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MAGIC-SAFE (Placebo Comparator): Parents will be provided with information about age-appropriate safety topics, including safe sleeping, car seats, baby-proofing, etc. The intervention is delivered via virtual visits, binder, website and newsletters.
  Interventions: Behavioral: MAGIC-SAFE
- MAGIC-FEED (Experimental): Parents will be provided with responsive feeding coaching to help them recognize hunger and satiety cues and nutrition coaching that includes bottle-/breast-feeding and complementary feeding in alignment with the Dietary Guidelines. The intervention is delivered via virtual visits, binder, website and newsletters.
  Interventions: Behavioral: MAGIC-FEED

INTERVENTIONS:
Behavioral: MAGIC-FEED — Parents will be provided with responsive feeding coaching to help them recognize hunger and satiety cues and nutrition coaching that includes bottle-/breast-feeding and complementary feeding in alignment with the Dietary Guidelines. The intervention is delivered via virtual visits, binder, website and newsletters.
  Arms: MAGIC-FEED
Behavioral: MAGIC-SAFE — Parents will be provided with information about age-appropriate safety topics, including safe sleeping, car seats, baby-proofing, etc. The intervention is delivered via virtual visits, binder, website and newsletters.
  Arms: MAGIC-SAFE

SUMMARY:
The study will use a longitudinal, randomized control trial design to determine intervention impact on parent and child behaviors, and infant health. The two intervention groups include: 1) MAGIC-FEED+; and 2) MAGIC-SAFE. This trial is an efficacy trial of the MAGIC-FEED and MAGIC-SAFE program that has been successfully implemented with families as part of the MAGIC 1.0 program trial (IRB#: 2015040017).

* The primary aim is to investigate each intervention's impact on infant BMIZ at 13 months.
* The investigators will also assess the effect of MAGIC-FEED on caregiver nutrition knowledge and feeding practices, responsive feeding, infant diet, and child self-regulatory abilities and assess how these factors impact child self-regulation of eating and adiposity.
* Finally, the investigators will determine if the interventions demonstrate the factors necessary to be a successful intervention as determined by the RE-AIM and PRISM frameworks.

DETAILED DESCRIPTION:
Obesity is a significant public health problem and risk begins early in life. In the US, over 19% of children ages 2-19 have obesity with 6% of these children classified with severe obesity. Obesity prevalence is lower among 2- to 5-year-old children (13.4%); however, by age 6, one in 5 children has obesity. Rapid weight gain over the first year of life is associated with overweight or obesity in toddlers and young children, which then tracks across the life course. It is critical to intervene on modifiable factors early in life to support healthy growth and prevent obesity. This trial is implemented across the first year in this population to support child diet quality, self-regulatory skills related to eating and growth to prevent obesity.

Interventions during the first year of life have been implemented to prevent child obesity. Most focus on breast and bottle feeding during the first 6 months or feeding across infancy. Few have demonstrated lasting effects beyond infancy on a relative body size measure that accounts for height such as BMIZ, and none have reported effects on long-term adiposity measured with a sensitive assessment tool or have successfully impacted long-term relative body size or adiposity. Further, prior RCTs have predominately been conducted via home visits. MAGIC 2.0 uses a virtual platform which will allows us to leverage the well-established effectiveness of home visiting to be accessible to caregivers with young children.

ELIGIBILITY:
Inclusion Criteria:

* A singleton infant 3-9 weeks of age, born ≥37 weeks gestation.
* The mother and other caregiver must be at least 18 years of age.
* The infant must live with the mother.
* Lives within the Austin metropolitan area.
* English or Spanish speaking.
* The primary caregiver must identify as the mother.

Exclusion Criteria:

* Infant diagnosed with major physical disabilities and/or medical condition that affects feeding and growth, and/or born <37 weeks gestation.
* Infant experienced NICU stay >7 days.
* Twins, triplets, or other multiples.
* Mothers and/or other caregivers younger than 18 years old.
* Mothers that do not consent to being video recorded with their baby.
* Families that do not speak either English or Spanish will be excluded from this study. Families that only speak English or Spanish, or families that speak English or Spanish and another language, will be accepted.
* Do not plan to remain in Austin area for the next two years.

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant Body Mass Index Z-score (BMIZ) at 13 and 24 months | 13 & 24 months
  Assessed via anthropometrics and WHO Child Growth Standards.
Infant dietary quality index | 0-13 months
  Infant dietary quality index (IDQI) score with higher scores indicating higher dietary quality (Au et al. J Nutr 2023, 153(3): 741-748). Calculated with questionnaire data from an adapted Infant Feeding Practices III Food Frequency Questionnaire.
Infant self-regulation during feeding | 0-13 months
  Infant self-regulation during feeding coded from video observation via the Nursing Child Assessment Feeding Scale.
Eating self-regulation | 24 months
  Assessed via 'Eating in the Absence of Hunger' experiment using standard protocols (Asta et al. Pediatrics 2016;137(5):e20153786).

SECONDARY OUTCOMES:
Caregiver nutrition knowledge | 0-24 months
  Caregiver nutrition knowledge assessed by the Infant Feeding Education Questionnaire.
Caregiver sensitivity | 0-24 months
  Caregiver responsive feeding/sensitivity with higher scores indicating greater sensitivity. Assessed by Chatoor's Feeding Scale, Hazen Sensitivity Scale and Nursing Child Assessment Feeding Scale.
Solid food introduction timing | 0-8 months
  Timing of solid food introduction (<6 mo, >=6 mo). Assessed by the adapted Infant Feeding Practices III Questionnaire.
Percentage body fat | 13 & 24 months
  Percentage body fat assessed via DXA.
Proportion with BMIZ >=95%ile | 13 & 24 months
  High BMI at 13 & 24 months
BMIZ change from 3 wk to 24 months | 0-24 months
  BMIZ change from 3 wk to 24 months assessed via anthropometrics and WHO Child Growth Standard.
Child self-regulation | 24 months
  Inhibitory control assessed via behavioral rating from the Barrier Box Tax with higher scores indicating greater regulation.
Caregiver infant feeding practices | 0-24 months
  Assessed by the Feeding Practices and Structure Questionnaire.
Baby Eating Behavior | ~ 8 months
  Infant eating behaviors assessed via the Baby Eating Behavior Questionnaire.
Child Eating Behavior | 24 months
  Child eating behaviors assessed via the Children's Eating Behavior Questionnaire.
Duration of exclusive breastfeeding | 0-24 months
  Duration of exclusive breastfeeding assessed via the adapted Infant Feeding Practices III Questionnaire.
Sugary beverages before 12 months | 0-12 months
  Introduction of sugary beverages prior to 12 months. Assessed via the adapted Infant Feeding Practices III questionnaire.
Child self-regulation | 13 months
  Assessed by the Brief Infant Toddler Social Emotional Assessment (BITSEA) with higher scores indicating greater self-regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Widen, PhD, RD, Principal Investigator — UT Austin; Deborah Jacobvitz, PhD, Principal Investigator — UT Austin
Locations (2):
- United States (2):
  - Sarah M. & Charles E. Seay Building, Austin, Texas
  - Dell Pediatric Research Institute, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided